CLINICAL TRIAL: NCT04477564
Title: Screening of Clonal Hematopoiesis of Indeterminate Potential in Venous Thromboembolism
Brief Title: Clonal Hematopoiesis of Indeterminate Potential in Venous Thromboembolism
Acronym: CHIPS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2020-01/SB-01
Record Dates: First submitted 2020-07-10; First posted 2020-07-20 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2023-06

CONDITIONS: Venous Thromboembolism
Keywords: Clonal Hematopoiesis of indeterminate potential
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — gDNA from leucocytes from a biobank (registration number DC-2008-290 and authorization number AC-2008-107)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Unprovoked proximal deep vein thrombosis
- Provoked distal deep vein thrombosis
- age-matched control group with no history of vein thrombosis

SUMMARY:
The aim of the study is to investigate the existence of clonal hematopoiesis of indeterminate potential (CHIP) in patients with a history of venous thromboembolism.

The study investigators make the assumption that these patients present mutations involved in CHIP occurrence.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 50 years old who have consulted at the Hematology laboratory of the Nîmes University Hospital for the occurrence or history of venous thromboembolism
* Patient who has accepted that their DNA was kept and used in the context of research on venous thromboembolism (biobank (registration number DC-2008-290 and authorization number AC-2008-107))

Exclusion Criteria:

* Patients less than 50 years old
* Patient who has refused that their DNA was kept and used in the context of research on venous thromboembolism

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women over 50 years old who have consulted at the Hematology laboratory of the Nîmes University Hospital for the occurrence or history of venous thromboembolism (Distal/proximal; Provoked/unprovoked) and who has accepted that their DNA was kept and used in the context of research on venous thromboembolism
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-07-03 (Actual); Primary Completion 2023-06-13 (Actual); Study Completion 2023-06-13 (Actual)

PRIMARY OUTCOMES:
DNMT3A mutations screening | For sequencing analysis: 2 months
  Next generation sequencing

SECONDARY OUTCOMES:
TET2, ASXL1, TP53, JAK2, SF3B1, SRSF2, GNB1, CBL, BCOR, SH2B3, PPM1D mutations screening | For sequencing analysis: 2 months
  Next generation sequencing

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nimes, Nîmes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Guillotin F, Mercier E, Fortier M, Bouvier S, Jacquet Q, Dallo M, Chea M, Bourguignon C, Cochery-Nouvellon E, Perez-Martin A, Gris JC. Clonal haematopoiesis of indeterminate potential in patients with venous thromboembolism. J Thromb Thrombolysis. 2023 Aug;56(2):351-354. doi: 10.1007/s11239-023-02836-4. Epub 2023 Jun 10. PMID 37300604